CLINICAL TRIAL: NCT03074435
Title: Insecticide Resistance Management in Burkina Faso and Côte D'Ivoire: Research on Vector Control Strategies
Brief Title: Insecticide Resistance Management in Burkina Faso and Côte D'Ivoire
Acronym: REACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Institut Pierre Richet (Other Government)
Responsible Party: Principal Investigator, Cédric PENNETIER, Principal Investigator, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: InstitutRD; 15SANIN213 (Other Grant/Funding Number: Expertise France)
Record Dates: First submitted 2016-11-04; First posted 2017-03-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Malaria
Keywords: Randomized Controlled Trials
MeSH Terms: conditions — Malaria | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized, parallel with baseline, trial. The study is bi-centric for the evaluation of two arms (LLIN+IRS and LLIN+BCC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control arm (LLIN-alone) (No Intervention): The baseline and control intervention (LLIN-alone) correspond to what is implemented in each country by their respective National Malaria Control Programs (NMCP). This include universal coverage with Long-Lasting insecticidal Nets (LLIN). This arm is common to both countries (Burkina Faso and Côte d'Ivoire)
- LLIN + indoor residual sprayings (Experimental): LLIN+IRS arm consisted in applying, in addition to LLINs, IRS with Actellic® 300CS (Syngenta AG, Basel, Switzerland) at a target dosage of 1 g. of active ingredient (pirimiphos-methyl) per m² in every houses of the selected villages. This arm is common to both countries (Burkina Faso and Côte d'Ivoire)
  Interventions: Device: Indoor residual sprayings
- LLIN + Larvicide (Experimental): The intervention consists in treating Anopheles breeding sites with BTI biological larvicide, in addition to LLINs. This arm was implemented in Côte d'Ivoire only.
  Interventions: Device: Larvicide
- LLIN+ One-health Ivermectin (Experimental): This arm consists in monthly injections of ivermectin to peri-domestic farm animals (mammals) during 4 consecutive months, oin addition to LLINs. This arm was implemented in Burkina Faso only.
  Interventions: Biological: Ivermectin
- LLIN + Behaviour Change Communication (Experimental): BCC complementary intervention (LLIN+BCC arm) was designed to target the following behaviors in the human population: (i) everyone sleep under an LLIN every night, (ii) every household and community member cleans up its environment to limits mosquito proliferation, (iii) every pregnant woman asks for, and takes the intermittent preventive treatment of malaria during pregnancy (ITP) and, (iv) people in charge of <5 y/o children come to see an health worker within 24h in case of fever. The intervention involve one health worker from the community per 35 households. Every health worker has the objective to perform 15 home visits (15-20 min), 20 interpersonal talks (15-20 min) and 4 group talks (15-30 min) per months.
  Interventions: Behavioral: BCC

INTERVENTIONS:
Device: Indoor residual sprayings — Houses will be spayed with this formulation containing Pyrimiphos methyl.
  Other Names: Actellic
  Arms: LLIN + indoor residual sprayings
Device: Larvicide — Larval breeding sites will be treated with larvicide
  Arms: LLIN + Larvicide
Behavioral: BCC
  Arms: LLIN + Behaviour Change Communication
Biological: Ivermectin
  Arms: LLIN+ One-health Ivermectin

SUMMARY:
This study evaluates the benefit to use 1) insecticide residual sprayings, 2) larvicides, 3) Ivermectin for domestic animals and 4) behaviour change communication strategy to complement the universal coverage with LLINs through a cluster randomized trial.

ELIGIBILITY:
For Cross-sectional surveys only, maximum age for participating in the study was 21 y/o in Côte d Ivoire and 18 y/o in Burkina Faso.

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15776 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Malaria incidence density | continuous monitoring during 2 years
  Malaria cases (whole population, every ages) registered in the local health system.

SECONDARY OUTCOMES:
Entomological Inoculation Rate | Every 8 weeks during 2 years
  Number of infectious bites/personn
Malaria prevalence | Every 4 months during 2 years
  % of positive blood smears among the 0-18 y/o population as recorded during cross sectional surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Pennetier, PhD, Principal Investigator — Institut de Rehcerche pour le Développement; Nicolas Moiroux, PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (2):
- Institut de Recherche en Sciences de la Santé, Bobo-Dioulasso, Burkina Faso
- Institut Pierre Richet, Bouaké, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bationo CS, Gaudart J, Dieng S, Cissoko M, Taconet P, Ouedraogo B, Some A, Zongo I, Soma DD, Tougri G, Dabire RK, Koffi A, Pennetier C, Moiroux N. Spatio-temporal analysis and prediction of malaria cases using remote sensing meteorological data in Diebougou health district, Burkina Faso, 2016-2017. Sci Rep. 2021 Oct 8;11(1):20027. doi: 10.1038/s41598-021-99457-9. PMID 34625589
- [Background] Taconet P, Porciani A, Soma DD, Mouline K, Simard F, Koffi AA, Pennetier C, Dabire RK, Mangeas M, Moiroux N. Data-driven and interpretable machine-learning modeling to explore the fine-scale environmental determinants of malaria vectors biting rates in rural Burkina Faso. Parasit Vectors. 2021 Jun 29;14(1):345. doi: 10.1186/s13071-021-04851-x. PMID 34187546
- [Background] Soma DD, Zogo B, Taconet P, Some A, Coulibaly S, Baba-Moussa L, Ouedraogo GA, Koffi A, Pennetier C, Dabire KR, Moiroux N. Quantifying and characterizing hourly human exposure to malaria vectors bites to address residual malaria transmission during dry and rainy seasons in rural Southwest Burkina Faso. BMC Public Health. 2021 Jan 30;21(1):251. doi: 10.1186/s12889-021-10304-y. PMID 33516197
- [Background] Soma DD, Zogo B, Hien DFS, Hien AS, Kabore DA, Kientega M, Ouedraogo AG, Pennetier C, Koffi AA, Moiroux N, Dabire RK. Insecticide resistance status of malaria vectors Anopheles gambiae (s.l.) of southwest Burkina Faso and residual efficacy of indoor residual spraying with microencapsulated pirimiphos-methyl insecticide. Parasit Vectors. 2021 Jan 18;14(1):58. doi: 10.1186/s13071-020-04563-8. PMID 33461621
- [Background] Soma DD, Zogo BM, Some A, Tchiekoi BN, Hien DFS, Pooda HS, Coulibaly S, Gnambani JE, Ouari A, Mouline K, Dahounto A, Ouedraogo GA, Fournet F, Koffi AA, Pennetier C, Moiroux N, Dabire RK. Anopheles bionomics, insecticide resistance and malaria transmission in southwest Burkina Faso: A pre-intervention study. PLoS One. 2020 Aug 3;15(8):e0236920. doi: 10.1371/journal.pone.0236920. eCollection 2020. PMID 32745085
- [Background] Zogo B, Soma DD, Tchiekoi BN, Some A, Ahoua Alou LP, Koffi AA, Fournet F, Dahounto A, Coulibaly B, Kande S, Dabire RK, Baba-Moussa L, Moiroux N, Pennetier C. Anopheles bionomics, insecticide resistance mechanisms, and malaria transmission in the Korhogo area, northern Cote d'Ivoire: a pre-intervention study. Parasite. 2019;26:40. doi: 10.1051/parasite/2019040. Epub 2019 Jul 12. PMID 31298995
- [Background] Zogo B, Koffi AA, Alou LPA, Fournet F, Dahounto A, Dabire RK, Baba-Moussa L, Moiroux N, Pennetier C. Identification and characterization of Anopheles spp. breeding habitats in the Korhogo area in northern Cote d'Ivoire: a study prior to a Bti-based larviciding intervention. Parasit Vectors. 2019 Mar 27;12(1):146. doi: 10.1186/s13071-019-3404-0. PMID 30917867
- [Background] Zogo B, Tchiekoi BN, Koffi AA, Dahounto A, Ahoua Alou LP, Dabire RK, Baba-Moussa L, Moiroux N, Pennetier C. Impact of sunlight exposure on the residual efficacy of biolarvicides Bacillus thuringiensis israelensis and Bacillus sphaericus against the main malaria vector, Anopheles gambiae. Malar J. 2019 Feb 26;18(1):55. doi: 10.1186/s12936-019-2687-0. PMID 30808348
- [Derived] Moiroux N, Zongo I, Assi SB, Some A, Tchiekoi NB, Zogo B, Soma DD, Hien DFDS, Taconet P, Ahoua Alou LP, Lefevre T, Cohuet A, Fournet F, Mouline K, Koffi AA, Dabire RK, Pennetier C. Efficacy of non-pyrethroid indoor residual spraying or intensive behaviour change communication in combination with long-lasting insecticidal nets for malaria control in west Africa: a pragmatic, cluster-randomised, controlled trial. Lancet Glob Health. 2025 Sep;13(9):e1605-e1616. doi: 10.1016/S2214-109X(25)00216-5. PMID 40845886